CLINICAL TRIAL: NCT04772118
Title: Improving Cancer Outcomes Through Personalized Care Planning and Symptom Managment
Brief Title: Improving Cancer Outcomes Through Personalized Care Planning and Symptom Management.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: G423 Multi TP
Record Dates: First submitted 2021-01-25; First posted 2021-02-26 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer; Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Carevive PROmpt™ — Patient Reported Outcomes Mobile Patient (Carevive PROmpt™), a digital cancer symptom monitoring platform.

SUMMARY:
This Study is a case control Study conducted with 100 patients with a solid tumor cancer diagnosis (lung, breast, or gynecologic cancer). Records of 50 patients who received treatment plans as standard of care will be abstracted for control data. 50 patients undergoing cancer treatment will receive a treatment plan and report symptoms using Carevive PROmPT™.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years of age or older.
* Subject participants must have a diagnosis of a breast, lung, or gynecologic cancer.
* Patients must have completed their navigation visit and received a Treatment Care Plan.
* Subjects must be able to complete on-line surveys using a cell phone, tablet, or computer.
* Subjects must be starting or receiving treatment.
* All participants must be able to understand English.

Exclusion Criteria:

* Any patient who cannot understand written or spoken English.
* Any patient without the ability to complete on-line surveys using a cell phone, tablet, or computer.
* Any prisoner and/or other vulnerable persons as defined by NIH (45 CFR 46, Subpart B, C and D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Outcomes for Primary Aim 1 - 50 intervention participants with a diagnosis for lung, breast or ovarian cancer measuring the prevalence and severity of 18 different symptoms reported from home over 3 months. | 10 months
  Aim 1 is to compare treatment side effect frequency and intensity and patient treatment adherence between Intervention and Control subjects.
  Data collection for this Aim includes side effect frequency and intensity and time on treatment. Patients in the intervention arm will complete the Core Assessment prior to enrollment as standard of care. They will be enrolled to use the Carevive PROmpt™ platform to access from home. Patients will be instructed to report symptoms once a week between clinic visits.
  Outcomes measures for this Aim are the prevalence and severity of symptoms in each group, adherence to symptom reporting from home in intervention participants, and time on treatment from enrollment to 3 months after enrollment.
  Prevalence will be determined by the number of symptom alerts per patient over 3 months/ Severity will be determined by the number of mild, moderate, severe, and very severe over 3 months.

SECONDARY OUTCOMES:
Outcomes for Secondary Aim 2 - 50 intervention patients will complete the Patient Satisfaction Survey at the 3month timepoint to measure satisfaction with treatment decision and care experience. | 10 months
  Aim 2 is to describe patient satisfaction with care experience and satisfaction with treatment decision.
  Patient satisfaction with care experience and satisfaction with treatment decision will be measured with the Patient Satisfaction Survey (Appendix E). This survey is derived from the Survey of Patient Experiences with Cancer Care Survey (i.e., the Cancer CAHPS) which was developed specifically for cancer patients and is used to evaluate satisfaction with care in the Oncology Care Model (OCM). Surveys will be completed by intervention patients at the three months visit (by paper or electronically) or from home (electronically or by phone administered by the RC) if no visit is planned.
Outcomes for Secondary Aim 3 - Feasibility will be measured by completion of the patient questionnaires and patient symptom reports by the 50 intervention patients. Usability will be measured through provider feedback. | 10 months
  Aim 3 is to determine feasibility/usability of the electronic treatment planning and symptom assessment for the intervention arm only.
  Feasibility will be determined by the number of patients enrolled compared to the number of patients approached, and of those declined the reasons for the decline.
  Usability will be determined by the results of the patient satisfaction survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Mitchell Cancer Institute, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No